CLINICAL TRIAL: NCT04687137
Title: Open-arm, Japan Expanded Access Program With Lanadelumab (TAK-743) for Japanese Patients With Hereditary Angioedema
Brief Title: Expanded Access Program With Lanadelumab for Japanese People With Hereditary Angioedema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-743-5007; U1111-1260-2704 (Other: WHO); jRCT2031200255 (Registry Identifier: jRCT)
Record Dates: First submitted 2020-12-03; First posted 2020-12-29 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — lanadelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TAK-743 (Experimental)
  Interventions: Drug: TAK-743 300 mg

INTERVENTIONS:
Drug: TAK-743 300 mg — TAK-743 300 mg, subcutaneous injection every 2 or 4 weeks
  Other Names: TAKHZYRO

SUMMARY:
The expanded access program allows people to gain access to an unlicensed treatment on compassionate grounds. Lanadelumab, also known as TAK-743, is a medicine to help prevent hereditary angioedema attacks. Lanadelumab is not yet licensed for use in Japan.

The main aim of this study is to allow Japanese teenagers and adults with type I or type II hereditary angioedema to be treated with lanadelumab, through the expanded access program in Japan.

Participants can either have taken part in the previous study SHP643-302 or can be new participants. Participants just completing study SHP643-302 who reach the criteria can automatically take part in this study. However, for new participants, the study doctor will check who can take part at the first study visit.

For those who can take part, new participants will receive injections of lanadelumab just under the skin. Eventually, after training, some of these will be able to inject themselves with lanadelumab in the same way. Participants who injected themselves with lanadelumab in study SHP643-302 can continue to do so during this study.

The study doctors will decide if each participant will be treated with lanadelumab every 2 weeks or every 4 weeks. Treatment with lanadelumab will continue until lanadelumab is commercially available in Japan or the sponsor (Takeda) stops the study.

Participants can visit the clinic during treatment if needed. If treatment continues after 6 months, participants will visit the clinic every 12 weeks for a check-up. This will include noting any hereditary angioedema attacks and side effects from the treatment. After 7 months of treatment, the study staff will check-up with each participant every 2 weeks by telephone.

After treatment has finished, participants will visit the clinic for a final-check-up 4 weeks later.

DETAILED DESCRIPTION:
This study is Japan Expanded Access Program with TAK-743. The study drug in this study is called TAK-743. TAK-743 will be administered to people who have Type I or II hereditary angioedema (HAE).

Two types of participants will be enrolled into this study:

* Participants who rollover from Study SHP643-302 (NCT04180163).
* Participants who are non-rollovers (ie, were not participants in Study SHP643-302).

Participants who discontinue from Study SHP643-302 after providing informed consent are not eligible to enroll in this study.

All participants will be asked to administer TAK-743 300 mg with subcutaneous injection every 2 weeks throughout this study. Participants who is stable with over 6-month administration of 300mg every 2 weeks can be switched to 300mg every 4 weeks.

This multi-center trial will be conducted in Japan (approximately 15 sites). The overall time to participate in this study is over 182 days. Participants will make multiple visits to the clinic basically every 2 weeks until Day 182, and will be contacted by telephone every 2 weeks after Day 182 plus multiple visit every 12 weeks after Day 182 for a follow-up assessment until study completion.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the Investigator, the participant is capable of understanding and complying with protocol requirements.
2. Be of Japanese descent, defined as born in Japan and having Japanese parents and Japanese maternal and paternal grandparents.
3. Male and female HAE participants who are 12 years of age or older at the time of screening.
4. Documented diagnosis of disease HAE (Type I or II) based on all of the following:

   * Documented clinical history consistent with HAE (subcutaneous [SC] or mucosal, nonpruritic swelling episodes without accompanying urticaria).
   * Diagnostic testing results obtained during screening (or a prior lanadelumab study) that confirm HAE Type I or II: C1-inhibitor (C1-INH) functional level <40% of the normal level. Participants with functional C1-INH level 40% to 50% of the normal level may be enrolled if they also have a C4 level below the normal range. Participants may be retested if results are incongruent with clinical history or believed by the Investigator to be confounded by long-term prophylaxis (LTP) use. It is understood that C1-INH therapy may alter the lab results of C1-INH assessments; therefore, the Investigator's discretion in collaboration with sponsor is advised for proper documentation of eligibility.
   * At least one of the following: Age at reported onset of first angioedema symptoms =<30 years, a family history consistent with HAE Type I or II, or C1q within normal range.
5. Non-rollover participants only: A historical baseline HAE attack rate of at least 1 attack per 4 weeks in the recent 1 year.
6. Rollover participants only: Participants from Study SHP643-302 are permitted to rollover and enroll into this study if:

   * They completed the treatment period of Study SHP643-302; and
   * They consented to enter Study TAK-743-5007 on or before Day 350 of the SHP643-302 study (since Day 378 of Study SHP643-302 is also Day 0 of Study TAK-743-5007, informed consent may be completed on Day 364 or this visit, if not already provided).
7. Adult participants and caregivers of subjects under the age of 20 are willing and able to read, understand, and sign an informed consent form. Participants aged 12 to 19, whose caregiver has provided informed consent, are willing and able to read, understand and sign an informed consent form (an assent form, if applicable) as much as possible.
8. Agree to adhere to the protocol-defined schedule of treatments, assessments, and procedures.
9. Males and females who are fertile and sexually active must adhere to contraception requirements for the duration of the study as follows:

   * Females of childbearing potential must agree to be abstinent or it is recommended to use highly effective forms of contraception from the screening period through 70 days after the final study visit.
   * Females of nonchildbearing potential, defined as surgically sterile (status post-hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or postmenopausal for at least 12 months do not require contraception during the study.
   * Males, including males who are surgically sterile (post-vasectomy), with female partners of childbearing potential must agree to be abstinent or else use a medically acceptable form of contraception from the screening period through 70 days after the final study visit.

Exclusion Criteria:

1. If rolling over from Study SHP643-302, presence of important safety concerns that would preclude participation in this study.
2. Concomitant diagnosis of another form of chronic, recurrent angioedema such as acquired angioedema, HAE with normal C1-INH (also known as HAE Type III/normal C1-INH), idiopathic angioedema, or recurrent angioedema associated with urticaria.
3. Dosing with an investigational drug (not including lanadelumab or other HAE therapies) or exposure to an investigational device within 4 weeks prior to screening.
4. Exposure to angiotensin-converting enzyme (ACE) inhibitors within 4 weeks prior to screening or any newly initiated or dose modification of estrogen-containing medications with systemic absorption (such as oral contraceptives or hormonal replacement therapy) 3 months prior to the screening visit.
5. Unwilling to discontinue short or long-term prophylactic therapy for HAE, eg, C1-INH, attenuated androgens or anti-fibrinolytics within 3 weeks after starting the treatment period. Short-term prophylaxis is defined as C1-INH, attenuated androgens, or antifibrinolytic used to avoid angioedema complications from medically indicated procedures.
6. Any of the following liver function test abnormalities: alanine aminotransferase (ALT) >3 × upper limit of normal (ULN), or aspartate aminotransferase (AST) >3 × ULN, or total bilirubin >2 × ULN (unless the bilirubin elevation is a result of Gilbert's syndrome).
7. Pregnancy or breast feeding.
8. Have any uncontrolled underlying medical condition which would require treatment adjustment during the study treatment period, that, in the opinion of the Investigator or sponsor, may confound the results of the safety assessments or may place the participant at risk. Participants with stable treatment for at least 3 months prior to screening and NOT expecting any change to their treatment regimen for 6 months during the study treatment period, will not be excluded.
9. Participant has a known hypersensitivity to the study drug or its components.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-06-18 (Actual); Study Completion 2022-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (9):
- Japan (9):
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Asahi General Hospital, Asahi, Chiba
  - Tomakomai City Hospital, Tomakomai, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Tokai University Hospital, Isehara, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Osaka University Hospital, Suita, Osaka
  - Saiyu Soka Hospital, Sōka, Saitama
  - Hiroshima University Hospital, Hiroshima

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5ff6fe77565ce300294c6abe

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 9 investigative centers in Japan from 10 February 2021 to 18 June 2022.
Pre-assignment Details: A total of 12 participants with type I and II hereditary angioderma (HAE) participated in this study. Two types of participants were enrolled into this study: Participants who rolled over from Study SHP643-302 (NCT04180163) and participants who were non-rollovers (i.e., were not participants in Study SHP643-302 [NCT04180163]).
Groups:
- Rollover Participants: Rollover participants from Study SHP643-302 (NCT04180163) in this group received lanadelumab 300 milligrams (mg) subcutaneous (SC) injection on Day 0 followed by every 2 weeks (q2w) or every 4 weeks (q4w) if well-controlled (attack-free) for 26 consecutive weeks with lanadelumab treatment based on Investigator's discretion.
- Non-rollover Participants: Non-rollover participants in this group received lanadelumab 300 mg SC on Day 0 followed by q2w or q4w if well-controlled (attack-free) for 26 consecutive weeks with lanadelumab treatment based on Investigator's discretion.
Period: Overall Study
Arm/Group | Rollover Participants | Non-rollover Participants
Started | 11 | 1
Completed | 11 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of study drug.
Groups:
- Rollover Participants: Rollover participants from Study SHP643-302 (NCT04180163) in this group received lanadelumab 300 mg SC injection on Day 0 followed by q2w or q4w if well-controlled (attack-free) for 26 consecutive weeks with lanadelumab treatment based on Investigator's discretion.
- Total: Total of all reporting groups
Arm/Group | Rollover Participants | Non-rollover Participants | Total
Number analyzed (Participants) | 11 | 1 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (12.56) | 41.0 | 42.3 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 9
  Male | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 1 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 1 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 11 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Including Serious TEAEs and Adverse Events of Special Interest (AESI)
Description: TEAEs were defined as adverse events (AEs) with onset at the time of or following the first exposure to lanadelumab in this study, or medical conditions present prior to the start of treatment but increasing in severity or relationship at the time of or following the start of treatment. Serious TEAEs were defined as any untoward clinical manifestation of signs, symptoms, outcomes (related to IP or not) that at any dose: resulted in death, was life-threatening, required inpatient/prolongation of hospitalization, resulted in persistent/significant disability/incapacity, congenital abnormality/birth defect, important medical event. AESI were defined as investigator-reported hypersensitivity reactions, events of disordered coagulation as bleeding/hypercoagulable. Relatedness to study drug was based on Investigator's discretion. TEAEs were classified and reported as Hereditary Angioedema (HAE) attack and non-HAE attack AEs in this outcome measure.
Time Frame: From start of study drug administration (in current study) up to end of study (EOS) (Day 294)
Population: FAS included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rollover Participants | Non-rollover Participants
Number analyzed (Participants) | 11 | 1
Participants
  Any TEAEs: Non-HAE | 11 | 1
  Any TEAEs: HAE | 8 | 1
  AESI: Non-HAE | 1 | 0
  AESI: HAE | 0 | 0
  Any Serious TEAEs: Non-HAE | 1 | 0
  Any Serious TEAEs: HAE | 1 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Tests
Description: Clinical laboratory testing included clinical serum chemistry, hematology, coagulation and urinalysis. Any change in clinical laboratory abnormalities which were deemed clinically significant by the investigator were recorded as TEAEs.
Time Frame: From start of study drug administration (in current study) up to EOS (Day 294)
Population: FAS included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rollover Participants | Non-rollover Participants
Number analyzed (Participants) | 11 | 1
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital signs parameters included blood pressure, heart rate, body temperature and respiratory rate. Any change in vital sign abnormalities which were deemed clinically significant by the investigator were recorded as TEAEs.
Time Frame: From start of study drug administration (in current study) up to EOS (Day 294)
Population: FAS included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rollover Participants | Non-rollover Participants
Number analyzed (Participants) | 11 | 1
Participants | 0 | 0

4. Secondary Outcome: Time to First HAE Attack After Day 0 for the Efficacy Evaluation Period for Non-Rollover Participants
Description: A HAE attack was defined as the symptoms or signs consistent with an attack in at least 1 of the following locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). The time to the first HAE attack (days) was calculated from the date and time of the first dose of lanadelumab for the efficacy evaluation period (Day 0 through Day 182) to the date and time of the first in HAE attack after the first open-label dose for the efficacy evaluation period of Day 0 through Day 182. The time to the first Investigator-confirmed HAE attack (days) was summarized using Kaplan-Meier (KM) methods.
Time Frame: Day 0 (in current study) through Day 182
Population: FAS included all participants who received at least 1 dose of study drug. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure. Data was not collected and analyzed for rollover participants as pre-specified in protocol.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Non-rollover Participants
Number analyzed (Participants) | 1
days | 0.0 [NA to NA] — 95% CI data could not be calculated as there are insufficient number of participants with event.

ADVERSE EVENTS:
Time Frame: From start of study drug administration (in current study) up to EOS (Day 294)
Description: FAS included all participants who received at least 1 dose of study drug.
Arm/Group | Rollover Participants | Non-rollover Participants
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/1
Other Adverse Events (participants affected / at risk) | 11/11 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rollover Participants (N=11) | Non-rollover Participants (N=1)
Hereditary angioedema (Congenital, familial and genetic disorders) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rollover Participants (N=11) | Non-rollover Participants (N=1)
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chillblains (Injury, poisoning and procedural complications) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Hereditary angioedema (Congenital, familial and genetic disorders) | 8 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Injection site erythema (General disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Myelopathy (Nervous system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Skin candida (Infections and infestations) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 4 | 1
Vaccination site pain (General disorders) | 1 | 0
Vaccination site swelling (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

.

DOCUMENTS (2):
  • Study Protocol (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT04687137/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT04687137/SAP_001.pdf